CLINICAL TRIAL: NCT07024420
Title: Effect of Sigh Ventilation on Postoperative Pulmonary Complications in Cardiac Surgery: A Multicenter, Randomized Controlled Trial
Brief Title: Sigh Ventilation in Cardiac Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Fengmei Guo, Deputy director, Zhongda Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SIVECS
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-09

CONDITIONS: Postoperative Pulmonary Complications (PPCs); Cardiac Surgery in Adult Patient
Keywords: Sigh Ventilation; Cardiac Surgery; Postoperative Pulmonary Complications

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sigh Ventilation (Experimental): sigh breaths, low tidal volume and moderate PEEP levels
  Interventions: Other: Sigh Breaths; Other: Low Tidal Volume; Other: Moderate PEEP
- Conventional Ventilation (Active Comparator): low tidal volume, moderate PEEP levels
  Interventions: Other: Low Tidal Volume; Other: Moderate PEEP

INTERVENTIONS:
Other: Sigh Breaths — Sigh breaths were added by elevating PEEP, targeting a plateau pressure of 35 cmH2O (or 40 cmH2O for patients with a Body Mass Index > 35 kg/m2). These sigh breaths were administered once every 6 minutes at predefined stages in the perioperative period from the time of anesthesia intubation until endotracheal extubation, postoperative day 7, or death, whichever occurred first, but not during transport. Each sigh consisted of the minimum number of respiratory cycles aimed to achieve a total duration of at least 5 seconds, based on the respiratory cycle duration preset on the ventilator.
  Arms: Sigh Ventilation
Other: Low Tidal Volume — 6-8ml/kg predicted body weight
Other: Moderate PEEP — PEEP set according to ARDSnet low PEEP- fraction of inspired oxygen table, FiO2 was set as the lowest fraction targeted to maintain SpO2 ≥ 96%

SUMMARY:
The purpose of this trial is to investigate whether sigh ventilation strategy, combining sigh breaths, low tidal volume, and moderate PEEP levels, protects against major pulmonary complications within the first 7 postoperative days after cardiac surgery, as compared with conventional ventilation strategy with low tidal volume, and moderate PEEP levels.

DETAILED DESCRIPTION:
Preventing postoperative pulmonary complications with the use of low tidal volume ventilation is now an established consensus. However, low tidal volume promote alveolar collapse in poorly ventilated, dependent regions of the lung.

Recruitment maneuvers, typically delivered at specific intraoperative timepoints, aimed to counteract alveolar collapse promoted by low tidal volume, was found to yield transient physiological benefits. And the PROVECS trial failed to show extra benefit of recruitment maneuvers in cardiac surgery patients in terms of pulmonary complications within the first 7 postoperative days, as compared with low tidal volume ventilation.

Sigh breaths, which involves cyclic deep inflations to re-expand alveoli, potentially providing sustained benefits. The purpose of this trial is to investigate the specific role of sigh breaths for reducing pulmonary complications in cardiac surgery patients already receiving protective ventilation with low tidal volume and moderate PEEP levels.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older;
* Elective cardiac surgery with cardiopulmonary bypass, aortic clamp and cardioplegia;
* Written informed consent is obtained from patients and/or their legal representatives.

Exclusion Criteria:

* Emergence surgery;
* Left ventricular assist device implantation;
* Planned thoracotomy with one lung ventilation;
* Undergo concurrent surgical procedures outside cardiology;
* Neuromuscular illness;
* Mechanical ventilation within the last 2 weeks before surgery, include CPAP and NIV;
* Preoperative shock;
* Preoperative Hypoxemia (PaO2<60mmHg OR SpO2<90% on ambient air);
* Preoperative left ventricular ejection fraction < 40%;
* Systolic pulmonary artery pressure > 50 mmHg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 686 (Estimated)
Dates: Start 2025-10-09 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of major postoperative pulmonary complications (Grade ≥ 3 ) through POD7 | From randomization to postoperative day 7
  Postoperative pulmonary complications were scored using a grade scale ranging from 0 to 5. Major postoperative pulmonary complications are defined as Grade ≥ 3.
  Grade 3 (Pleural effusion, pneumonia, pneumothorax, HFNC OR NIV support, re-intubation), Grade 4 (IMV dependence ≥ 48h, HFNC OR NIV dependence ≥ 48h ), Grade 5 (Death).

SECONDARY OUTCOMES:
Severity of postoperative pulmonary complications through POD7 | From randomization to postoperative day 7
  Postoperative pulmonary complications were scored using a grade scale ranging from 0 to 5. Using the worst score within POD7 for analysis.
  Grade 0 (No symptom of interest), Grade 1 (Dry cough, microatelectasis, dyspnea), Grade 2 (Productive cough, bronchospasm, hypoxemia, atelectasis, hypercarbia), Grade 3 (Pleural effusion, pneumonia, pneumothorax, HFNC OR NIV support, re-intubation), Grade 4 (IMV dependence ≥ 48h, HFNC OR NIV dependence ≥ 48h ), Grade 5 (Death).
Proportion of major postoperative pulmonary complications (Grade ≥ 3 ) through hospitalization | From randomization up to hospital discharge, assessed up to postoperative day 30
  Postoperative pulmonary complications were scored using a grade scale ranging from 0 to 5. Major postoperative pulmonary complications are defined as Grade ≥ 3.
  Grade 3 (Pleural effusion, pneumonia, pneumothorax, HFNC OR NIV support, re-intubation), Grade 4 (IMV dependence ≥ 48h, HFNC OR NIV dependence ≥ 48h ), Grade 5 (Death).
Severity of postoperative pulmonary complications through hospitalization | From randomization up to hospital discharge, assessed up to postoperative day 30
  Postoperative pulmonary complications were scored using a grade scale ranging from 0 to 5. Using the worst score within hospitalization for analysis.
  Grade 0 (No symptom of interest), Grade 1 (Dry cough, microatelectasis, dyspnea), Grade 2 (Productive cough, bronchospasm, hypoxemia, atelectasis, hypercarbia), Grade 3 (Pleural effusion, pneumonia, pneumothorax, HFNC OR NIV support, re-intubation), Grade 4 (IMV dependence ≥ 48h, HFNC OR NIV dependence ≥ 48h ), Grade 5 (Death).
No Ventilatory Support Days by POD7 | From randomization to postoperative day 7
  Days alive and not receive IMV, HFNC, and NIV support
No Ventilatory Support Days by POD30 | From randomization to postoperative day 30
  Days alive and not receive IMV, HFNC, and NIV support
Proportion of Acute Respiratory Distress Syndrome through hospitalization | From randomization up to hospital discharge, assessed up to postoperative day 30
  ARDS diagnosed according to the 2023 ATS New Global Definition
Intensive Care Unit length of stay by POD30 | From randomization to postoperative day 30
Hospital length of stay by POD30 | From randomization to postoperative day 30
30-day mortality | From randomization to postoperative day 30
  The proportion of patients who died within postoperative day 30

OTHER OUTCOMES:
Shock-free days | From randomization to postoperative day 30
  Shock was defined as receiving any intravenous infusion of vasopressor/inotropic (i.e. norepinephrine, epinephrine, phenylephrine, vasopressin analogues, angiotensin, dopamine, dobutamine, milrinone or levosimendan), and patients transferred out of the ICU were assumed to be shock free. A value of 0 free days for patients who died before POD30.
Barotrauma | From randomization up to hospital discharge, assessed up to postoperative day 30
  Barotrauma includes pneumothorax, pneumomediastinum, or subcutaneous emphysema.
Pneumothorax | From randomization up to hospital discharge, assessed up to postoperative day 30
  Pneumothorax detected through chest X-ray or CT scan
New-onset atrial fibrillation | From randomization to hospital discharge, assessed up to postoperative day 30
  New-onset atrial fibrillation detected through ECG
Ventricular fibrillation | From randomization to hospital discharge, assessed up to postoperative day 30
  Ventricular fibrillation detected through ECG
Cardiac arrest | From randomization to hospital discharge, assessed up to postoperative day 30
  The proportion of patients with cardiac arrest
Other adverse events | From randomization to hospital discharge, assessed up to postoperative day 30
  The proportion of other adverse events related to the interventions assessed by investigators

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda Hospital, Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Study data without patient information
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Related papers published 3 months later, the IPD will be shared
Access Criteria: fmguo2022@163.com , wang15zc@163.com

REFERENCES:
- [Result] Lagier D, Velly LJ, Guinard B, Bruder N, Guidon C, Vidal Melo MF, Alessi MC. Perioperative Open-lung Approach, Regional Ventilation, and Lung Injury in Cardiac Surgery. Anesthesiology. 2020 Nov 1;133(5):1029-1045. doi: 10.1097/ALN.0000000000003539. PMID 32902561
- [Result] Lagier D, Fischer F, Fornier W, Huynh TM, Cholley B, Guinard B, Heger B, Quintana G, Villacorta J, Gaillat F, Gomert R, Degirmenci S, Colson P, Lalande M, Benkouiten S, Minh TH, Pozzi M, Collart F, Latremouille C, Vidal Melo MF, Velly LJ, Jaber S, Fellahi JL, Baumstarck K, Guidon C; PROVECS Study Group. Effect of open-lung vs conventional perioperative ventilation strategies on postoperative pulmonary complications after on-pump cardiac surgery: the PROVECS randomized clinical trial. Intensive Care Med. 2019 Oct;45(10):1401-1412. doi: 10.1007/s00134-019-05741-8. Epub 2019 Oct 1. PMID 31576435